CLINICAL TRIAL: NCT05068505
Title: Effectiveness of a Community Health Worker Delivered Care Intervention for Hypertension Control in Uganda: a Stepped Wedge, Cluster Randomized Control Trial
Brief Title: Effectiveness of a Community Health Worker Delivered Care Intervention for Hypertension Control in Uganda
Acronym: CHW-HTC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: University of Miami (Other); Makerere University (Other); Yale University (Other); London School of Hygiene and Tropical Medicine (Other); Johns Hopkins University (Other); Ministry of Health, Uganda (Other Government); African Community Center for Social Sustainability (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. med. Felix Knauf, Director of the Charité Mitte Campus - Senior Physician, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: Balamu2021
Record Dates: First submitted 2021-09-15; First posted 2021-10-06 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Hypertension; Community Health Workers
Keywords: Hypertension; Community health workers; Uncontrolled blood pressure; Uganda
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participant Recruiters
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community health worker delivered multicomponent intervention (Experimental): The study will employ a closed cohort stepped wedge cluster randomized design. There will be a sequential crossover of clusters from the control to the intervention arms and the order of the cross over will be randomly determined. This study will be conducted in 21 clusters within Nakaseke district. Each cluster will consist of 4-5 villages. We plan to rollout the intervention in three clusters per month.
  Interventions: Behavioral: Community health worker delivered multicomponent intervention
- Control (No Intervention): All clusters will be observed under both the intervention and control arm through sequential crossover.

INTERVENTIONS:
Behavioral: Community health worker delivered multicomponent intervention — The multi-component intervention will be centered on monthly household visits by trained CHWs for a period of seven months in a rural setting in Nakaseke, Uganda, consisting of the following; (1) blood pressure and sugar monitoring; (2) BMI monitoring; (3) cardiovascular disease risk assessment; (4) Using checklists to guide monitoring and referral to clinics; (5) healthy lifestyle counselling and education. During home visits, CHWs will remind patients of follow-up visits. We will measure blood pressure at baseline and 3-monthly for the entire cohort. We will conduct individual-level mixed effects analyses of study data, adjusting for time and clustering by patient and community.
  We will conduct an interim analysis at 3 months to assess differences between groups. If a statistically significant difference is detected the intervention will be applied across the remaining clusters
  Arms: Community health worker delivered multicomponent intervention

SUMMARY:
Over 80% of the morbidity and mortality related to non-communicable diseases (NCDs) occurs in low-income and middle-income countries (LMICs). Community health workers (CHWs) may improve disease control and medication adherence among patients with NCDs in LMICs, but data are scarce, particularly in sub-Saharan African settings. In Uganda, and the majority of LMICs, management of uncontrolled blood pressure remains limited in constrained health systems. Intervening at the primary care level, using CHWs to improve medical treatment outcomes has not been well studied. The investigators aim to determine the effectiveness of a CHW-led intervention in blood pressure control among confirmed hypertensive patients and patient-related factors associated with uncontrolled hypertension. Methods: Conduction of a stepped-wedge cluster randomized controlled trial study of 869 adult patients with hypertension attending two NCD clinics to test the effectiveness, acceptability and fidelity of a CHW-led intervention. The multi-component intervention will be centered on monthly household visits by trained CHWs for a period of seven months, consisting of the following; (1) blood pressure and sugar monitoring; (2) BMI monitoring; (3) cardiovascular disease risk assessment; (4) Using checklists to guide monitoring and referral to clinics; (5) healthy lifestyle counselling and education. During home visits, CHWs will remind patients of follow-up visits. The investigators will measure blood pressure at baseline and 3-monthly for the entire cohort. The investigators will additionally test acceptability of the intervention and fidelity over the course of the intervention. The investigators will conduct individual-level mixed effects analyses of study data, adjusting for time and clustering by patient and community. Conclusion: The results of this study will inform community delivered hypertension management across a range of LMIC settings.

ELIGIBILITY:
Inclusion Criteria:

* Participants with hypertension (Systolic >140 and/or Diastolic >90)
* Participants attending the two NCD clinics
* Adults 18 years and above
* Participants residing in the three sub counties (Nakaseke Town Council, Nakaseke Sub County and Kasangombe of Nakaseke district)
* Participants able to give informed consent.

Exclusion Criteria:

* Patients diagnosed with hypertension but already controlled
* Pregnant women
* Patients with an expected life expectancy of less than one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 869 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Blood pressure control | 3 months
  Decrease in the average systolic and/or diastolic blood pressure between the intervention and control arms.

SECONDARY OUTCOMES:
Glycemic control | 3 months
  Defined as a reduction >1% in heamoglobin A1C
Proportion of participants with blood pressure control | 3 months
  Defined as blood pressure <140/90 mmHg

OTHER OUTCOMES:
Composite negative clinical cardiovascular disease (CVD) outcomes | 3 months
  Including CVD related admissions, stroke, and myocardial infarction, incident heart failure will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Felix Knauf, Prof.Dr.med., Principal Investigator — Charité University, Berlin, Germany
Locations (1):
- Makerere University College of Health Sciences, Kampala, Uganda

REFERENCES:
- [Derived] Ingenhoff R, Nandawula J, Siddharthan T, Ssekitoleko I, Munana R, Bodnar BE, Weswa I, Kirenga BJ, Mutungi G, van der Giet M, Kalyesubula R, Knauf F. Effectiveness of a community health worker-delivered care intervention for hypertension control in Uganda: study protocol for a stepped wedge, cluster randomized control trial. Trials. 2022 May 24;23(1):440. doi: 10.1186/s13063-022-06403-9. PMID 35610712